CLINICAL TRIAL: NCT02755467
Title: A Clinical Evaluation of the Treatment of Spider Angioma Using a Dual Wavelength Laser Emitting 532 nm Laser Energy
Brief Title: Clinical Evaluation of the Treatment of Spider Angioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EV08
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Spider Angioma
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser treatment (Experimental): Each subject will receive a 532 nm KTP laser treatment for their spider angioma(s).
  Interventions: Device: KTP laser

INTERVENTIONS:
Device: KTP laser — Dual Wavelength Laser Emitting 532 nm Laser Energy
  Other Names: Cutera Excel V

SUMMARY:
To evaluate the safety and effectiveness of the laser treatment for the treatment of spider angiomas.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the 532 nm KTP laser within the Cutera Excel V system for the treatment of spider angiomas.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 5 to 65 years of age (inclusive).
2. Fitzpatrick Skin Types I-IV
3. Subject must be able to read, understand and sign the Informed Consent Form.
4. If subject is a minor (<18 years old in Illinois), Assent must be obtained from the subject and a Parental Consent Form must be signed by the parents or legal guardian.
5. Subject must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
6. Willing to have limited sun exposure for the duration of the study, including the follow-up period.
7. Willingness to have digital photographs taken of their spider angioma(s) and agree to use of photographs for presentation, educational or marketing purposes
8. Agree not to undergo any other procedure for the treatment of spider angioma during the study.

Exclusion Criteria:

1. Pregnant.
2. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
3. Having a known anti-coagulative condition or taking anticoagulation medications, including aspirin.
4. History of seizure disorders due to light.
5. Systemic use of isotretinoin (Accutane®) within 6 months of study participation.
6. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
7. Participation in a study of another device or drug within 3 months prior to enrollment or during the study.
8. In the opinion of the investigator, any physical or mental condition which might make it unsafe for the subject to participate in this study or which requires systemic therapy that could interfere with this research study.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Stankiewicz, MD FAAD, Principal Investigator — DuPage Medical Group
Locations (1):
- DuPage Medical Group, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Treatment
Started | 22
Completed | 21
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Laser Treatment
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Physician's Global Assessment Scale for Improvement of Spider Angioma
Description: Assessment of Baseline vs. 4 weeks post-final treatment for improvement of spider angiomas using the Physician's Global Assessment scale.
  High scores indicate better outcomes:
  0. None
  1. Mild
  2. Moderate
  3. Significant
  4. Very Significant
  5. Complete Removal
Time Frame: Four weeks post laser treatment.
Population: 1 subject was lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Laser Treatment
Number analyzed (Participants) | 21
score on a scale | 4.5 (0.6)

ADVERSE EVENTS:
Time Frame: 4 weeks post final laser treatment
Arm/Group | Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 14/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatment (N=22)
Erythema (Skin and subcutaneous tissue disorders) | 9
Purpura (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No